CLINICAL TRIAL: NCT03590899
Title: Semi-manual Vessel Density Analysis on Optical Coherence Tomography Angiography Images of Healthy Adults
Status: Completed | Type: Observational
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Miklos Schneider MD, PhD, Principal Investigator, Assistant Professor of Ophthalmology, Head of General Outpatient Unit, Semmelweis University
Other Study IDs: VESDEN-OCTA-1253
Record Dates: First submitted 2018-06-13; First posted 2018-07-18 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Healthy patients: Healthy volunteers without retinal disease, glaucoma, previous ocular surgery, laser photocoagulation, or optical media opacities that would disturb imaging.
  Interventions: Device: Optical coherence tomography angiography (Zeiss Cirrus HD OCT 5000 AngioPlex)

INTERVENTIONS:
Device: Optical coherence tomography angiography (Zeiss Cirrus HD OCT 5000 AngioPlex) — Non-invasive, non-contact optical coherence tomography angiography scans of the retina are done per built-in device protocol using the Zeiss Cirrus HD OCT 5000 AngioPlex machine.

SUMMARY:
Purpose of the study is to examine the vessel density of healthy adults' optical coherence tomography angiography images with two semi-manual methods and an automated quantification program.

DETAILED DESCRIPTION:
Optical coherence tomography angiography (OCTA) is a software upgrade on conventional spectral-domain or swept-source optical coherence tomography devices that enables non-invasive, dye-free, three dimensional analysis of the retinal vessels.

Vessel density is a very important parameter almost in all retinal disorders. In the recent past, automated quantification software was built into some OCTA devices which can automatically calculate the retinal vessel density as well.

In this study two semi-manual techniques are used in order to analyze the vessel density of healthy subjects' OCTA images. Vessel density is also measured with a new automated quantification program, and results of the three methods are compared.

OCT machines are approved in the EU and the US and are not experimental devices.

The device used in this study is the commercially available Zeiss Cirrus HD OCT Angioplex 5000 that operates with spectral-domain technology.

ELIGIBILITY:
Inclusion Criteria:

* healthy patients without eye disease

Exclusion Criteria:

* incapacity
* any history or clinical evidence of retinal disease or glaucoma
* previous ocular surgery or laser photocoagulation
* optical media opacities that would disturb imaging

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: White Caucasian
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Vessel density (VD) measured by Mexican Hat filtering technique | Through study completion, 1 year
  Following standard OCTA imaging with Zeiss Cirrus Angioplex, images are transferred to ImageJ and proportion of the vessels and the total image area (white pixels2/total number of pixels2) is calculated using Mexican Hat filtering technique.
Skeleton density (SD) measured by Mexican Hat filtering technique | Through study completion, 1 year
  Following standard OCTA imaging with Zeiss Cirrus Angioplex, images are transferred to ImageJ and length of blood vessels (white skeletonized pixels/total number of pixels2) is calculated using Mexican Hat filtering technique.
Vessel diameter index (VDI) measured by Mexican Hat filtering technique | Through study completion, 1 year
  Represents the average vessel caliber (two dimensional white pixels in the binarized image/one dimensional white pixels in the skeletonized image or VD/SD) using Mexican Hat filtering technique.
Vessel density (VD) measured by Shanbag tresholding technique | Through study completion, 1 year
  Following standard OCTA imaging with Zeiss Cirrus Angioplex, images are transferred to ImageJ and proportion of the vessels and the total image area (white pixels2/total number of pixels2) is calculated using Shanbag tresholding technique.
Skeleton density (SD) measured by Shanbag tresholding technique | Through study completion, 1 year
  Following standard OCTA imaging with Zeiss Cirrus Angioplex, images are transferred to ImageJ and length of blood vessels (white skeletonized pixels/total number of pixels2) is calculated using Shanbag tresholding technique.
Vessel diameter index (VDI) measured by Shanbag tresholding technique | Through study completion, 1 year
  Represents the average vessel caliber (two dimensional white pixels in the binarized image/one dimensional white pixels in the skeletonized image or VD/SD) using Shanbag tresholding technique.
Vessel density (VD) measured by Angioplex Metrix | Through study completion, 1 year
  Following standard OCTA imaging with Zeiss Cirrus Angioplex measurement is done by built-in non-disclosed VD algorithm owned by Zeiss.
Skeleton density (SD) measured by Angioplex Metrix | Through study completion, 1 year
  Following standard OCTA imaging with Zeiss Cirrus Angioplex measurement done by built-in non-disclosed SD algorithm owned by Zeiss.

SECONDARY OUTCOMES:
Comparison of results obtained by the three quantification techniques | Through study completion, 1 year
  Comparison of VD and SD (see above) obtained by Mexican Hat filtering technique, Shanbag tresholding technique and built-in Zeiss proprietary algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Miklós Schneider, MD, PhD, Principal Investigator — Semmelweis University, Department of Ophthalmology
Locations (1):
- Semmelweis University, Department of Ophthalmology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spaide RF, Klancnik JM Jr, Cooney MJ. Retinal vascular layers imaged by fluorescein angiography and optical coherence tomography angiography. JAMA Ophthalmol. 2015 Jan;133(1):45-50. doi: 10.1001/jamaophthalmol.2014.3616. PMID 25317632
- [Background] Kashani AH, Chen CL, Gahm JK, Zheng F, Richter GM, Rosenfeld PJ, Shi Y, Wang RK. Optical coherence tomography angiography: A comprehensive review of current methods and clinical applications. Prog Retin Eye Res. 2017 Sep;60:66-100. doi: 10.1016/j.preteyeres.2017.07.002. Epub 2017 Jul 29. PMID 28760677
- [Background] Coscas F, Sellam A, Glacet-Bernard A, Jung C, Goudot M, Miere A, Souied EH. Normative Data for Vascular Density in Superficial and Deep Capillary Plexuses of Healthy Adults Assessed by Optical Coherence Tomography Angiography. Invest Ophthalmol Vis Sci. 2016 Jul 1;57(9):OCT211-23. doi: 10.1167/iovs.15-18793. PMID 27409475
- [Background] Corvi F, Pellegrini M, Erba S, Cozzi M, Staurenghi G, Giani A. Reproducibility of Vessel Density, Fractal Dimension, and Foveal Avascular Zone Using 7 Different Optical Coherence Tomography Angiography Devices. Am J Ophthalmol. 2018 Feb;186:25-31. doi: 10.1016/j.ajo.2017.11.011. Epub 2017 Nov 21. PMID 29169882
- [Background] Matsunaga D, Yi J, Puliafito CA, Kashani AH. OCT angiography in healthy human subjects. Ophthalmic Surg Lasers Imaging Retina. 2014 Nov-Dec;45(6):510-5. doi: 10.3928/23258160-20141118-04. PMID 25423629
- [Background] Tan PE, Balaratnasingam C, Xu J, Mammo Z, Han SX, Mackenzie P, Kirker AW, Albiani D, Merkur AB, Sarunic MV, Yu DY. Quantitative Comparison of Retinal Capillary Images Derived By Speckle Variance Optical Coherence Tomography With Histology. Invest Ophthalmol Vis Sci. 2015 Jun;56(6):3989-96. doi: 10.1167/iovs.14-15879. PMID 26098464
- [Background] Lupidi M, Coscas F, Cagini C, Fiore T, Spaccini E, Fruttini D, Coscas G. Automated Quantitative Analysis of Retinal Microvasculature in Normal Eyes on Optical Coherence Tomography Angiography. Am J Ophthalmol. 2016 Sep;169:9-23. doi: 10.1016/j.ajo.2016.06.008. Epub 2016 Jun 11. PMID 27296485
- [Background] Weinhaus RS, Burke JM, Delori FC, Snodderly DM. Comparison of fluorescein angiography with microvascular anatomy of macaque retinas. Exp Eye Res. 1995 Jul;61(1):1-16. doi: 10.1016/s0014-4835(95)80053-0. PMID 7556462
- [Background] Mendis KR, Balaratnasingam C, Yu P, Barry CJ, McAllister IL, Cringle SJ, Yu DY. Correlation of histologic and clinical images to determine the diagnostic value of fluorescein angiography for studying retinal capillary detail. Invest Ophthalmol Vis Sci. 2010 Nov;51(11):5864-9. doi: 10.1167/iovs.10-5333. Epub 2010 May 26. PMID 20505200
- [Background] Agrawal R, Xin W, Keane PA, Chhablani J, Agarwal A. Optical coherence tomography angiography: a non-invasive tool to image end-arterial system. Expert Rev Med Devices. 2016 Jun;13(6):519-21. doi: 10.1080/17434440.2016.1186540. Epub 2016 May 25. No abstract available. PMID 27176114
- [Background] Munk MR, Giannakaki-Zimmermann H, Berger L, Huf W, Ebneter A, Wolf S, Zinkernagel MS. OCT-angiography: A qualitative and quantitative comparison of 4 OCT-A devices. PLoS One. 2017 May 10;12(5):e0177059. doi: 10.1371/journal.pone.0177059. eCollection 2017. PMID 28489918
- [Background] Zudaire E, Gambardella L, Kurcz C, Vermeren S. A computational tool for quantitative analysis of vascular networks. PLoS One. 2011;6(11):e27385. doi: 10.1371/journal.pone.0027385. Epub 2011 Nov 16. PMID 22110636
- [Background] Reif R, Qin J, An L, Zhi Z, Dziennis S, Wang R. Quantifying optical microangiography images obtained from a spectral domain optical coherence tomography system. Int J Biomed Imaging. 2012;2012:509783. doi: 10.1155/2012/509783. Epub 2012 Jun 26. PMID 22792084
- [Background] De Vitis LA, Benatti L, Tomasso L, Baldin G, Carnevali A, Querques L, Querques G, Bandello F. Comparison of the Performance of Two Different Spectral-Domain Optical Coherence Tomography Angiography Devices in Clinical Practice. Ophthalmic Res. 2016;56(3):155-62. doi: 10.1159/000447094. Epub 2016 Jul 12. PMID 27399271
- [Background] Shin JW, Sung KR, Lee JY, Kwon J, Seong M. Optical coherence tomography angiography vessel density mapping at various retinal layers in healthy and normal tension glaucoma eyes. Graefes Arch Clin Exp Ophthalmol. 2017 Jun;255(6):1193-1202. doi: 10.1007/s00417-017-3671-4. Epub 2017 Apr 20. PMID 28429123
- [Background] Choi J, Kwon J, Shin JW, Lee J, Lee S, Kook MS. Quantitative optical coherence tomography angiography of macular vascular structure and foveal avascular zone in glaucoma. PLoS One. 2017 Sep 21;12(9):e0184948. doi: 10.1371/journal.pone.0184948. eCollection 2017. PMID 28934255
- [Background] Gadde SG, Anegondi N, Bhanushali D, Chidambara L, Yadav NK, Khurana A, Sinha Roy A. Quantification of Vessel Density in Retinal Optical Coherence Tomography Angiography Images Using Local Fractal Dimension. Invest Ophthalmol Vis Sci. 2016 Jan 1;57(1):246-52. doi: 10.1167/iovs.15-18287. PMID 26803800
- [Background] Al-Sheikh M, Ghasemi Falavarjani K, Akil H, Sadda SR. Impact of image quality on OCT angiography based quantitative measurements. Int J Retina Vitreous. 2017 May 15;3:13. doi: 10.1186/s40942-017-0068-9. eCollection 2017. PMID 28515959
- [Background] Schneider CA, Rasband WS, Eliceiri KW. NIH Image to ImageJ: 25 years of image analysis. Nat Methods. 2012 Jul;9(7):671-5. doi: 10.1038/nmeth.2089. PMID 22930834
- [Background] Kim AY, Chu Z, Shahidzadeh A, Wang RK, Puliafito CA, Kashani AH. Quantifying Microvascular Density and Morphology in Diabetic Retinopathy Using Spectral-Domain Optical Coherence Tomography Angiography. Invest Ophthalmol Vis Sci. 2016 Jul 1;57(9):OCT362-70. doi: 10.1167/iovs.15-18904. PMID 27409494